CLINICAL TRIAL: NCT06104254
Title: Determining the Effect of Preoperative Education on Orthopedic Surgery Patients on Pain Beliefs and Pain-Related Care Needs in the Postoperative Period
Brief Title: Education Importance and Pain Belief Differences Among Patients Who Underwent Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ismailasatir
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Orthopedic Disorder; Post Operative Pain
Keywords: post operative pain; pain beliefs; patient education
MeSH Terms: conditions — Musculoskeletal Diseases; Pain, Postoperative | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): The patient who assign to control group, they will give standard ward care before surgery and we measure their pain beliefs and pain level. After operation we will asses their pain beliefs and pain level. the last measure will be carried out after 30 days operation.
- experimental group (Experimental): The patient who assign to experimental group, we will measure their pain beliefs and pain level before surgery. After that a researcher will give an education before operation to these patients about pain, potential pain and pain management after surgery. we will asses these patients pain beliefs and pain level after surgery and 30 days later again.
  Interventions: Other: education

INTERVENTIONS:
Other: education — we will give an education to experimental group about pain and pain management.
  Arms: experimental group

SUMMARY:
The assessment of pain plays a crucial role in pain management. Nurses are instrumental in the identification, evaluation, and initiation of pain management strategies. In the literature, it is strongly recommended to provide education about postoperative pain management to patients, their families, and those responsible for patient care. Additionally, the development of a pain management plan and goals is advocated.

The optimal timing, content, and objectives of patient education depend on the type of pain (acute or chronic), the availability and effectiveness of treatment, and the patient's level of education and literacy. Educating individuals undergoing elective surgery or outpatient treatment about the likelihood and magnitude of acute pain they may experience, as well as informing them about available methods to prevent or alleviate this pain, is critical for pain management. Shindo et al. conducted a study suggesting that perioperative pain education significantly reduces postoperative opioid use.

According to the Health Belief Model, an individual's perception of health is influenced by their perception of the value of health, beliefs about illness, and beliefs about the consequences of illness. Therefore, when a patient's health beliefs and attitudes are determined, health education and treatment planning can be tailored more appropriately.

DETAILED DESCRIPTION:
The assessment of pain plays a crucial role in pain management. Nurses are instrumental in the identification, evaluation, and initiation of pain management strategies. In the literature, it is strongly recommended to provide education about postoperative pain management to patients, their families, and those responsible for patient care. Additionally, the development of a pain management plan and goals is advocated.

The optimal timing, content, and objectives of patient education depend on the type of pain (acute or chronic), the availability and effectiveness of treatment, and the patient's level of education and literacy. Educating individuals undergoing elective surgery or outpatient treatment about the likelihood and magnitude of acute pain they may experience, as well as informing them about available methods to prevent or alleviate this pain, is critical for pain management. Shindo et al. conducted a study suggesting that perioperative pain education significantly reduces postoperative opioid use.

According to the Health Belief Model, an individual's perception of health is influenced by their perception of the value of health, beliefs about illness, and beliefs about the consequences of illness. Therefore, when a patient's health beliefs and attitudes are determined, health education and treatment planning can be tailored more appropriately.

Preoperative education is a significant component of the surgical process. Preoperative patient education is known to contribute to reduced postoperative pain and anxiety, as well as early discharge. Grä Sjöling et al. (2003) demonstrated in their study that preoperative education/information had an impact on postoperative pain scores. Furthermore, another study indicated that the majority of patients' greatest concern was the pain they might experience in the postoperative period. The information provided to patients about pain is associated with a high level of satisfaction. In this study, the aim is to determine the beliefs about postoperative pain and pain scores of patients undergoing orthopedic surgery following preoperative education. In this context, the study also aims to highlight the importance of involving patients in pain management and the preoperative patient education in the literature.

In this regard, the objective of the study is to examine the effects of postoperative mobilization times on patients' recovery status, pain levels, quality of life, and the development of complications after spinal surgery. By reporting the results of the study, it is anticipated that contributions will be made to the literature and that it will serve as a source for future research.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years old.
* being conscious
* there have not any auditory and understanding problem
* being an elective surgery patient

Exclusion Criteria:

* Being under 18 years of age,
* being unconscious,
* Rheumatoid arthritis patients,
* Patients with mental illness,
* Patients using psychiatric drugs,
* Patients with a known history of cancer
* Patients requiring urgent surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Pain level | before operation and after surgery in the 30 days process
  we will use to measure patient pain level Numeric Pain Scale (NPS) several times. The intensity of pain will measure the area in which the individual mark between 0 (no pain) and 10 (worst pain i felt in my life).
Pain Beliefs | before operation and after surgery in the 30 days process
  we will use to measure patient' pain belief with Pain Beliefs Questionnaire. Edwards and coworkers developed this survey to measure patients' pain beliefs in 1992. the survey has 12 questions. Likert-type scale items range from 1. (never) to 6 (always). An increase in the score obtained from the scale sub-dimension indicates a high pain belief in the sub-dimension, and a decrease in the score indicates a low pain belief in the relevant sub-dimension. Thanks to this survey we can measure both psychological and organic pain beliefs of patients. we will use the survey several times in different stages.

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University Faculty of Health Science, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No